CLINICAL TRIAL: NCT05460039
Title: Technology-mediated Dance: Impact on Psychossocial, Physical, and Cognitive Functions of the Old
Brief Title: Impact of a Technology Mediated Dance Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aveiro University (Other)
Responsible Party: Principal Investigator, Anabela G Silva, Assistant Professor, Aveiro University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DanceMove
Record Dates: First submitted 2022-07-14; First posted 2022-07-15 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Older Adults Without Any Specific Clinical Condition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual activities (No Intervention): This group will receive no intervention.
- DanceMove (Experimental): This group will perform dance sessions mediated by technology (a dance mat and a web platform).
  Interventions: Other: Dance mediated by tecnhology

INTERVENTIONS:
Other: Dance mediated by tecnhology — A web system and a dance mat are used to stimulate participants to perform dance activities for 8 weeks.
  Arms: DanceMove

SUMMARY:
This study aims to investigate whether a technology-mediated dance impacts on psychosocial, physical and cognitive functions of the old adults when compared to usual activities.

DETAILED DESCRIPTION:
This study aims to investigate whether a technology-mediated dance impacts on psychosocial, physical, and cognitive functions of old adults when compared to usual activities. It will have two arms one of which will receive a dance mat and perform dance sessions for 8 weeks, while the other group will continue their usual activities. Participants will be assessed for psychosocial, physical, and cognitive aspects at baseline, end of the intervention, and at 3 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* People living independently in the community
* 65 years old or older
* With no cognitive impairment defined based on the 6-item cognitive decline test [4]
* Independent at walking without walking aids
* Access to a personal computer and internet
* For older adults unable to use a computer, a patient or carer with digital literacy needs to be identified for the older adult to enter the study.

Exclusion Criteria:

* Reporting cardiovascular pathology that limits the performance of the dance or dizziness or imbalance prior to using the mat

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Gait velocity | Baseline
  Assessed using the gait velocity test, i.e., the velocity of gait when walking in a straight line for 4 meters; it is measured in meters per second.
Gait velocity | After the intervention (8 weeks after baseline assessment)
  Assessed using the gait velocity test, i.e., the velocity of gait when walking in a straight line for 4 meters; it is measured in meters per second.
Gait velocity | At 3 months follow up
  Assessed using the gait velocity test, i.e., the velocity of gait when walking in a straight line for 4 meters; it is measured in meters per second.

SECONDARY OUTCOMES:
Balance | Baseline
  Balance will be assessed through the Functional Reach Test, which measures the ability of a person to reach forward without moving the feet; it is measured in cm.
Balance | After the intervention (8 weeks after baseline assessment)
  Balance will be assessed through the Functional Reach Test, which measures the ability of a person to reach forward without moving the feet; it is measured in cm.
Balance | At 3 months follow up
  Balance will be assessed through the Functional Reach Test, which measures the ability of a person to reach forward without moving the feet; it is measured in cm.
Cognitive functioning | Baseline
  This will be measured using the Trail Making Test which is a paper-based test; score is given in seconds.
Cognitive functioning | After the intervention (8 weeks after baseline assessment)
  This will be measured using the Trail Making Test which is a paper-based test; score is given in seconds.
Cognitive functioning | At 3 months follow up
  This will be measured using the Trail Making Test which is a paper-based test; score is given in seconds.
Pain intensity | Baseline
  Measured with a 100 mm Vertical Numeric Pain Rating Scale, anchored with 0 (no pain) and 100 (worst possible pain)
Pain intensity | After the intervention (8 weeks after baseline assessment)
  Measured with a 100 mm Vertical Numeric Pain Rating Scale, anchored with 0 (no pain) and 100 (worst possible pain)
Pain intensity | At 3 months follow up
  Measured with a 100 mm Vertical Numeric Pain Rating Scale, anchored with 0 (no pain) and 100 (worst possible pain)
Quality of life | Baseline
  Measured using the WHOQOL-Bref (WHO Quality of Life questionnaire); scores range between 0 to 20 and higher scores indicate better quality of life
Quality of life | After the intervention (8 weeks after baseline assessment)
  Measured using the WHOQOL-Bref (WHO Quality of Life questionnaire); scores range between 0 to 20 and higher scores indicate better quality of life
Quality of life | At 3 months follow up
  Measured using the WHOQOL-Bref (WHO Quality of Life questionnaire); scores range between 0 to 20 and higher scores indicate better quality of life
Health status | Baseline
  Measured using the EuroQoL EQ-5D; scores range from 5 to 25 and higher scores; indicate lower quality of life (note: according to the EuroQol Research Foundation, EQ-5D is not an abbreviation and is the correct term to use in print or verbally)
Health status | After the intervention (8 weeks after baseline assessment)
  Measured using the EuroQoL EQ-5D; scores range from 5 to 25 and higher scores; indicate lower quality of life (note: according to the EuroQol Research Foundation, EQ-5D is not an abbreviation and is the correct term to use in print or verbally)
Health status | At 3 months follow up
  Measured using the EuroQoL EQ-5D; scores range from 5 to 25 and higher scores; indicate lower quality of life (note: according to the EuroQol Research Foundation, EQ-5D is not an abbreviation and is the correct term to use in print or verbally)
Self-efficacy | Baseline
  Measured using the Perceived Self-Efficacy Scale; scores vary between 10 and 40 and higher scores indicate higher self-efficacy
Self-efficacy | After the intervention (8 weeks after baseline assessment)
  Measured using the Perceived Self-Efficacy Scale; scores vary between 10 and 40 and higher scores indicate higher self-efficacy
Self-efficacy | At 3 months follow up
  Measured using the Perceived Self-Efficacy Scale; scores vary between 10 and 40 and higher scores indicate higher self-efficacy
Loneliness | Baseline
  Measured using the University of California, Los Angeles, Loneliness Scale; scores vary between 4 and 28 and higher scores indicate higher loneliness
Loneliness | After the intervention (8 weeks after baseline assessment)
  Measured using the University of California, Los Angeles, Loneliness Scale; scores vary between 4 and 28 and higher scores indicate higher loneliness
Loneliness | At 3 months follow up
  Measured using the University of California, Los Angeles, Loneliness Scale; scores vary between 4 and 28 and higher scores indicate higher loneliness
Social support | Baseline
  Measured with the Oslo Social Support Scale (OSSS-3) with Life Events Scale; score varies between 3 and 14 and higher scores indicate stronger social support
Social support | After the intervention (8 weeks after baseline assessment)
  Measured with the Oslo Social Support Scale (OSSS-3) with Life Events Scale; score varies between 3 and 14 and higher scores indicate stronger social support
Social support | At 3 months follow up
  Measured with the Oslo Social Support Scale (OSSS-3) with Life Events Scale; score varies between 3 and 14 and higher scores indicate stronger social support

CONTACTS AND LOCATIONS:
Overall Officials: Anabela Silva, Principal Investigator — School of Health Sciences, University of Aveiro
Locations (1):
- School of Health Sciences, Aveiro, Portugal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silva AG, Martins AI, Andias R, Nery E, Silva T, Ribeiro O, Santinha G, Rocha NP. A web step-based digital solution's impact on physical, cognitive and psychosocial functioning of community-dwelling older adults: A mixed methods randomized and controlled trial. Internet Interv. 2024 Aug 21;38:100766. doi: 10.1016/j.invent.2024.100766. eCollection 2024 Dec. PMID 39280041